CLINICAL TRIAL: NCT04882891
Title: Holter of Movement in Patients with Multiple Sclerosis. Acti-SEP Study: Uncontrolled Environment.
Brief Title: Holter of Movement in Patients with Multiple Sclerosis in Uncontrolled Environment.
Acronym: ActiMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: SYSNAV (Industry); Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Laurent Servais, Professor, Centre Hospitalier Universitaire de Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ActiMS - uncontrolled
Record Dates: First submitted 2021-03-11; First posted 2021-05-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: Actimyo; Accelerometry; Home monitoring
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: all patients undergo clinical evaluation and wear Actimyo device in daily living to assess their gait and its evolution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MS patients (Experimental): Ambulant patients with multiple sclerosis
  Interventions: Device: Actimyo

INTERVENTIONS:
Device: Actimyo — Actimyo° is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.

SUMMARY:
ActiSEP is a multicentric academic study. Ambulant patients with multiple sclerosis may be included on a voluntary basis. The investigators plan to include a group of approximately 80 patients with MS, fulfilling the McDonald's 2017 criteria, of whom 40 of them show a progressive course according to the Lublin classification.

The investigators have planned two visits (at baseline and 1 year later). On both visits, participants will perform few tests (timed 25-Foot Walk (T25-FW), 9-Hole Peg Test (9-HPG), 6-minutes walk test (6MWT), Berg balance scale) and will answer to some questionaires (Godin Leisure Time Exercice Questionnaire, multiple sclerosis walking scale, modified fatigue impact scale, Hospital Anxiety and Depression Scale) After each visit, participants will wear Actimyo for three months in daily living.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MS diagnosis,
* Over 18 years old,
* Ambulant patients,
* Signed informed consent,
* No clinical and / or radiological relapse within 3 months.
* EDSS < or = à 5,5,
* Treated patient must be on a stable regimen dose and molecule for at least 2 month prior to inclusion.

Exclusion Criteria:

* Patients with excessive cognitive disorders, limiting the understanding of task or with apparent communication difficulties hindering data collection.
* Any other previous or present pathology having an impact on motor function.
* Recent surgery or trauma (less than 6 months) in the upper or lower limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
95th centile of stride velocity | 1 year
  95th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter per second).
50th centile of stride velocity | 1 year
  50th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter per second).
95th centile of stride length | 1 year
  95th centile of stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).
50th centile of stride length | 1 year
  50th centile of stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).
Stance phase time | 1 year
  Stance time over full stride time for each foot obtained with a magneto-inertial sensor (Actimyo°) in real-life (percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Poleur, MD, Principal Investigator — CHR Citadelle-CHU liège
Locations (7):
- Belgium (5):
  - Centre Hospitalier Universitaire de Liège, Liège, Liège
  - CHR Citadelle, Liège, Liège
  - Antwerp University Hospital, Antwerp
  - CHC Mont Legia, Liège
  - Saint-Luc University Clinics, Woluwe-St. Lambert
- France (2):
  - Hôpital d'instruction des Armées Percy, Clamart
  - Pitié-Salpêtrière Hospital, Paris

IPD SHARING:
Plan to Share IPD: No